CLINICAL TRIAL: NCT02191865
Title: Pharmacokinetics, Safety and Tolerability of Nintedanib Single Oral Dose in Male and Female Patients With Different Degrees of Hepatic Impairment (Child-Pugh Classification A and B) as Compared With Nintedanib Administration to Male and Female Healthy Subjects (a Non-blinded, Parallel Group Study of Phase I)
Brief Title: Nintedanib in Volunteers With Hepatic Impairment Compared With Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.200; 2014-000690-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — nintedanib

ARMS (3):
- Mild liver impairment (Experimental): Patients with mild hepatic impaired function (Child-Pugh A)
  Interventions: Drug: Nintedanib
- Moderate liver impairment (Experimental): Patients with moderate hepatic impaired function (Child-Pugh B)
  Interventions: Drug: Nintedanib
- Healthy volunteers (Experimental): Healthy control subjects
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Soft gelatine capsule
  Arms: Moderate liver impairment
Drug: Nintedanib — Soft gelatine capsule
  Arms: Mild liver impairment
Drug: Nintedanib — Soft gelatine capsule
  Arms: Healthy volunteers

SUMMARY:
The primary objective of this study is to investigate the effect of mild (Child-Pugh A, score 5-6) and moderate (Child-Pugh B, score 7-9) hepatic impairment on the pharmacokinetics, safety and tolerability of nintedanib, in comparison with a control group with normal hepatic function following oral administration of nintedanib as single dose.

ELIGIBILITY:
Inclusion criteria:

Healthy subjects:

* Male or female subject, healthy according to the investigator's judgement based on a complete medical history, including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory
* Age of 18 to 79 years at screening visit

Hepatically impaired patients as determined by a hepatologist/ gastroenterologist:

* A documented diagnosis of the impaired hepatic function, determined by hepatologist/gastroenterologist/specialist for internal medicine, must be available in the patient´s source data.
* Male or female chronic hepatically impaired patient as determined by screening results and classified as Child-Pugh A (Child-Pugh score of 5-6 points) or as Child-Pugh B (Child-Pugh score of 7-9 points). Hepatic insufficiency must be diagnosed at least 3 months before screening.
* Age of 18 to 79 years at screening visit

Exclusion criteria:

Healthy subjects:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range at screening visit that the investigator considers to be of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders judged as clinically relevant by the investigator
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication based on the investigator´s judgment
* Women who are breast feeding or of child-bearing potential not using a highly effective method of birth control for at least one month prior to inclusion and at least 3 month after administration of trial medication.

Hepatically impaired patients as determined by a hepatologist/gastroenterologist:

* Medical disorder, condition or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Patients with significant diseases other than underlying diagnose of hepatic impairment and concomitant diseases related to it. A significant disease is defined as a disease which in the opinion of the investigator:

  * put the patient at risk because of participation in the study
  * may influence the results of the study
  * is not in a stable condition
* Surgery of the gastrointestinal tract that could interfere with the kinetics of the trial medication based on the investigator´s judgment
* Women who are breast feeding or of child-bearing potential not using a highly effective method of birth control for at least one month prior to inclusion and at least 3 month after administration of trial medication

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1199.200.49001 Boehringer Ingelheim Investigational Site, Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were to be matched to subjects with hepatic impairment ((Child-Pugh A, score 5 or 6),(Child-Pugh B, score 7 to 9)) by age (±10 years), body weight (±10%), sex, race, and smoking habits (current vs. ex- and never smokers).
Groups:
- Child Pugh A: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with mild hepatic impairment (Child-Pugh A).
  Subjects were dosed in a 3 plus 5 design, where a subgroup of 3 subjects was dosed and safety was evaluated formally at a safety meeting prior to dosing the remaining 5 subjects in the group.
- Child Pugh B: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with moderate hepatic impairment (Child-Pugh B).
  Subjects were dosed in a 3 plus 5 design, where a subgroup of 3 subjects was dosed and safety was evaluated formally at a safety meeting prior to dosing the remaining 5 subjects in the group.
- Healthy: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in subjects with normal hepatic function.
Period: Overall Study
Arm/Group | Child Pugh A | Child Pugh B | Healthy
Started | 8 | 8 | 17
Completed | 8 | 8 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set (TS) included all subjects who were dispensed study medication and were documented to have taken atleast one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Child Pugh A | Child Pugh B | Healthy | Total
Number analyzed (Participants) | 8 | 8 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.1) | 56.6 (6.5) | 57.6 (8.4) | 58.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 13
  Male | 5 | 5 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-inf) of Nintedanib
Description: AUC (0-inf) (Area under the concentration-time curve of the Nintedanib in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: Pre-dose and 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h and 168h after drug administration
Population: Pharmacokinetic set (PKS): The PKS included all subjects of the TS who provided at least 1 observation for at least 1 primary PK endpoint, which was judged as PK evaluable and was not affected by important protocol violation(s) relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Child-Pugh A: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with mild hepatic impairment (Child-Pugh A).
- Child-Pugh B: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with moderate hepatic impairment (Child-Pugh B).
- Healthy Matched Child-Pugh A: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in healthy control subjects matched with hepatic (Child pugh A) impaired subjects
- Healthy Matched Child-Pugh B: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in healthy control subjects matched with hepatic (Child pugh B) impaired subjects .
Arm/Group | Child-Pugh A | Child-Pugh B | Healthy Matched Child-Pugh A | Healthy Matched Child-Pugh B
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 200 (87.7) | 674 (66.3) | 92.7 (58.5) | 77.8 (38.2)
Statistical Analysis 1: Comparison: Child-Pugh A vs Healthy Matched Child-Pugh A; The statistical model used for the analysis of AUC (0-inf) was an ANOVA (analysis of variance) model on the logarithmic scale. Observations from a subject with hepatic impairment and the matched healthy control subject were analysed as a matched pair; Test type: Superiority or Other; ANOVA; Fixed effect: 'hepatic status'; indicated whether a subject with hepatic impairment or a healthy subject , Random effect: 'matched pair'; ratio of the geometric means = 215.39, 90% CI 2-sided [120.71 to 384.32], Standard Deviation 73.5 — Ratio of Child Pugh A (Test): Healthy Child Pugh A (Reference). The Standard deviation is the Intra-individual gCV
Statistical Analysis 2: Comparison: Child-Pugh B vs Healthy Matched Child-Pugh B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 867.13, 90% CI 2-sided [572.93 to 1312.41], Standard Deviation 45.9 — Ratio of Child Pugh B (Test): Healthy Child Pugh B (Reference). The Standard deviation is the Intra-individual gCV

2. Primary Outcome: Cmax of Nintedanib
Description: Cmax (Maximum measured concentration of the Nintedanib in plasma)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Child-Pugh B: Oral administration of 1 soft gelatin capsule of 100 mg Nintedanib with 240 ml of water under fed conditions in patients with moderate hepatic impairment (Child-Pugh B).
Arm/Group | Child-Pugh A | Child-Pugh B | Healthy Matched Child-Pugh A | Healthy Matched Child-Pugh B
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 20.5 (68.4) | 59.4 (87.0) | 9.25 (54.1) | 7.81 (49.3)
Statistical Analysis 1: Comparison: Child-Pugh A vs Healthy Matched Child-Pugh A; The statistical model used for the analysis of Cmax was an ANOVA (analysis of variance) model on the logarithmic scale. Observations from a subject with hepatic impairment and the matched healthy control subject were analysed as a matched pair; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the geometric means = 221.76, 90% CI 2-sided [134.73 to 365.01], Standard Deviation 61.4 — Ratio of Child Pugh A (Test): Healthy Child Pugh A (Reference). The Standard deviation is the Intra-individual gCV
Statistical Analysis 2: Comparison: Child-Pugh B vs Healthy Matched Child-Pugh B; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 761.01, 90% CI 2-sided [439.01 to 1319.18], Standard Deviation 69.1 — Ratio of Child Pugh B (Test): Healthy Child Pugh B (Reference). The Standard deviation is the Intra-individual gCV

3. Secondary Outcome: AUC (0-tz) of Nintedanib
Description: AUC (0-tz) (Area under the concentration-time curve of the Nintedanib in plasma over the time interval from 0 to the last quantifiable drug plasma concentration)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Child-Pugh A | Child-Pugh B | Healthy Matched Child-Pugh A | Healthy Matched Child-Pugh B
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 193 (89.5) | 652 (66.2) | 89.2 (59.6) | 74.8 (38.9)
Statistical Analysis 1: Comparison: Child-Pugh A vs Healthy Matched Child-Pugh A; The statistical model used for the analysis of AUC (0-tz) was an ANOVA (analysis of variance) model on the logarithmic scale. Observations from a subject with hepatic impairment and the matched healthy control subject were analysed as a matched pair; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of the geometric means = 216.79, 90% CI 2-sided [120.37 to 390.45], Standard Deviation 75.0 — Ratio of Child Pugh A (Test): Healthy Child Pugh A (Reference). The Standard deviation is the Intra-individual gCV
Statistical Analysis 2: Comparison: Child-Pugh B vs Healthy Matched Child-Pugh B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 870.74, 90% CI 2-sided [576.36 to 1315.49], Standard Deviation 45.7 — Ratio of Child Pugh B (Test): Healthy Child Pugh B (Reference). The Standard deviation is the Intra-individual gCV

4. Secondary Outcome: Number (%) of Subjects With Drug-related Adverse Events (AEs)
Description: Number (%) of subjects with drug-related Adverse events (AEs)
Time Frame: (AEs) during the 'on-treatment' period (from administration of trial medication until the end of the 28-day residual effect period); Up to 29 days
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Child-Pugh A | Child-Pugh B | Healthy
Number analyzed (Participants) | 8 | 8 | 17
percentage of participants | 0.0 | 37.5 | 17.6

ADVERSE EVENTS:
Time Frame: AEs during the 'on-treatment' period (from administration of trial medication until the end of the 28-day residual effect period); up to 29 days
Groups:
- Child Pugh A: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with mild hepatic impairment (Child-Pugh A).
- Child Pugh B: Oral administration of 1 soft gelatin capsule of Nintedanib 100 mg with 240 ml of water under fed conditions in patients with moderate hepatic impairment (Child-Pugh B).
Arm/Group | Child Pugh A | Child Pugh B | Healthy
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/17
Other Adverse Events (participants affected / at risk) | 0/8 | 3/8 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Child Pugh A (N=8) | Child Pugh B (N=8) | Healthy (N=17)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights